CLINICAL TRIAL: NCT03508869
Title: Mirvaso® Gel and Dysport® for Erythema and Flushing of Rosacea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: sponsor asked site to suspend study.
Sponsor: Skin Laser & Surgery Specialists (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, David J. Goldberg, MD, Principal Investigator, Skin Laser & Surgery Specialists
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MG-DYS-ROS
Record Dates: First submitted 2016-05-19; First posted 2018-04-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Erythema and Flushing Associated With Rosacea
MeSH Terms: conditions — Erythema | interventions — Brimonidine Tartrate; Gels; abobotulinumtoxinA

ARMS (3):
- Mirvaso® (brimonidine) topical gel, 0.33% (Active Comparator): Mirvaso® (brimonidine) topical gel, 0.33% is an alpha adrenergic agonist indicated for the topical treatment of persistent facial erythema of rosacea in adults 18 years of age or older.
  Interventions: Drug: Mirvaso® (brimonidine) topical gel, 0.33%
- Dysport® (Active Comparator): Dysport® is an acetylcholine release inhibitor and a neuromuscular blocking agent.
  Interventions: Drug: Dysport®
- Dysport® in conjunction with Mirvaso (Active Comparator): Dysport® in conjunction with Mirvaso
  Interventions: Drug: Dysport® in conjunction with Mirvaso (brimonidine) topical gel, 0.33%

INTERVENTIONS:
Drug: Mirvaso® (brimonidine) topical gel, 0.33% — Mirvaso® (brimonidine) topical gel, 0.33% is an alpha adrenergic agonist indicated for the topical treatment of persistent facial erythema of rosacea in adults 18 years of age or older.
  Arms: Mirvaso® (brimonidine) topical gel, 0.33%
Drug: Dysport® — Dysport® is an acetylcholine release inhibitor and a neuromuscular blocking agent.
  Other Names: Dysport® (abobotulinumtoxinA)
  Arms: Dysport®
Drug: Dysport® in conjunction with Mirvaso (brimonidine) topical gel, 0.33% — Dysport® in conjunction with Mirvaso (brimonidine) topical gel, 0.33%
  Arms: Dysport® in conjunction with Mirvaso

SUMMARY:
To evaluate the safety and efficacy of Mirvaso® Gel and Dysport® for erythema and flushing of Rosacea.

DETAILED DESCRIPTION:
To assess the improvement of facial erythema and flushing while using Mirvaso® and Dysport® treatments based on the clinician's and patient's assessments using a verified 5-point grading scale

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. 18 years of age or older
3. Clinical diagnosis of rosacea
4. Moderate to severe persistent facial erythema associated with rosacea at baseline, as determined by: a grade of greater than or equal to 3 on the 5 point grading scale1 (Figure 1)
5. No known medical conditions that may interfere with study participation
6. Willingness to not use any products on their face for the duration of the study
7. Read, understand, and sign informed consent forms
8. Willingness to sign photography release form
9. Willing and able to comply with all follow-up requirements
10. Willingness to undergo treatment using Mirvaso® Gel and Dysport®

Exclusion Criteria:

1. Any significant skin disease at treatment area
2. Any medical condition which could interfere with the treatment
3. Inability or unwillingness to follow the treatment schedule
4. Inability or unwillingness to sign the informed consent
5. Pregnant or lactating
6. Allergy to cow's milk protein
7. Previous or current use of Mirvaso® Gel
8. Known hypersensitivity to Dysport® , Mirvaso® Gel or any of their ingredients
9. Previous Dysport® treatment 6 months prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Efficacy Assessments for Erythema | 6 months
  % of subjects who achieve a grade of 0 or 1 on the 5-point grading scale for Erythema 6 months post Dysport treatment Subject achieving a grade of 0 or 1 or ≥ 2 grade of improvement from baseline at 6 months for Erythema on the 5-point grading scale.
Efficacy Assessments for Flushing | 6 months
  % of subjects who achieve a grade of 0 or 1 on the 5-point grading scale for Flushing 6 months post Dysport treatment Subject achieving a grade of 0 or 1 or ≥ 2 grade of improvement from baseline at 6 months for Flushing on the 5-point grading scale.

SECONDARY OUTCOMES:
Safety Assessments | 6 months
  Safety evaluations will be performed at all visits. Adverse events, local tolerability (dryness, pruritus burning/stinging) and a facial exam will be performed for all visits.